CLINICAL TRIAL: NCT03780673
Title: Efficacy of the Combination of Simvastatin Plus Rifaximin in Patients With Decompensated Cirrhosis to Prevent ACLF Development: a Multicenter, Double-blind, Placebo Controlled Randomized Clinical Trial
Brief Title: Efficacy of the Combination of Simvastatin Plus Rifaximin in Patients With Decompensated Cirrhosis to Prevent ACLF Development
Acronym: 2018-001698-25
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Judit Pich (Other)
Responsible Party: Sponsor-Investigator, Judit Pich, Clinical Research Manager. CTU Clinic, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Organization: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIVERHOPE_EFFICACY
Record Dates: First submitted 2018-11-29; First posted 2018-12-19 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Liver Cirrhoses
MeSH Terms: interventions — Simvastatin; Rifaximin

STUDY DESIGN:
Intervention Model Description: Phase III, multicentre, double-blind placebo-controlled, randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: Neither the participants nor the researchers will know which group the participants has been allocated to
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simvastatin 20 mg + Rifaximin 400 mg (Experimental): Simvastatin 20 mg/day and rifaximin 400 mg/8 hours orally for 12 months
  Interventions: Drug: Simvastatin; Drug: Rifaximin
- Placebo of Simvastatin + Placebo of Rifaximin (Placebo Comparator): Placebo of simvastatin and placebo of rifaximin orally for 12 months
  Interventions: Drug: Placebo of Simvastatin; Drug: Placebo of Rifaximin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 20 mg/day for 12 months
  Arms: Simvastatin 20 mg + Rifaximin 400 mg
Drug: Rifaximin — Rifaximin 400/8 hours for 12 months
  Arms: Simvastatin 20 mg + Rifaximin 400 mg
Drug: Placebo of Simvastatin — Placebo of Simvastatin once a day for 12 months
  Arms: Placebo of Simvastatin + Placebo of Rifaximin
Drug: Placebo of Rifaximin — Placebo of Rifaximin/8 hours for 12 months
  Arms: Placebo of Simvastatin + Placebo of Rifaximin

SUMMARY:
The aim of this study is to assess the efficacy of oral administration of simvastatin plus rifaximin in patients with decompensated cirrhosis to halt the progression of the disease as assessed by prevention of the development of ACLF

DETAILED DESCRIPTION:
The current study was aimed at assessing whether a treatment based on combination of rifaximin and simvastatin would be effective in patients with decompensated cirrhosis to prevent ACLF development Considering that statins have been scarcely investigated in patients with decompensated cirrhosis due to a concern of potential higher liver and muscle toxicity in this population, a first LIVERHOPE_SAFETY clinical trial (unpublished) was undergone to assess safety and toxicity of statins with decompensated cirrhosis.

As a preliminary result of the LIVERHOPE_SAFETY clinical trial, it was concluded that the dose of Simvastatin 20mg per day plus Rifaximin is not associated to a higher risk of liver or muscle toxicity in patients with decompensated cirrhosis and simvastatin 20 mg was established for the LIVERHOPE_EFFICACY study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Cirrhosis defined by standard clinical criteria, ultrasonographic findings and/or histology
* Child-Pugh patients or Child-Pugh C patients (up to 12 points)
* Women of child-bearing potential must have a negative pregnancy test in serum before the inclusion in the study and agree to use highly effective contraceptive methods during the study. Highly effective contraceptive methods will include: intrauterine device, bilateral tubal occlusion, vasectomized partner and sexual abstinence.

Exclusion Criteria:

* Patients on treatment with statins or rifaximin up to one month before study inclusion.
* Patients with contraindications for statins or rifaximin therapy.
* Known hypersensitivity to simvastatin or rifaximin (or rifamycin derivatives).
* Patients with CK elevation of 50% or more above the upper limit of normal at study inclusion.
* Patients on treatment with potent inhibitors of CYP3A4 enzyme
* Patients on treatment with drugs with potential interactions with simvastatin
* Patients with previous history of myopathy.
* Patients with previous history of intestinal obstruction or those who are at increased risk of this complication.
* Patients with ACLF according to the criteria published by Moreau et al.
* Serum creatinine ≥2 mg/dL (176.8 μmol/L).
* Serum bilirubin>5 mg/dL (85.5 μmol/L).
* 12. INR ≥2.5
* Bacterial infection within 10 days before study inclusion.
* Gastrointestinal bleeding within 10 days before study inclusion.
* Current overt hepatic encephalopathy, defined as grade II-IV hepatic encephalopathy according to the New-Haven classification.
* Patients with active hepatocellular carcinoma or history of hepatocellular carcinoma that is in remission for less than six months for uninodular HCC or for less than 12 months for multinodular HCC within Milan criteria.
* Patients on antiviral therapy for HCV or those who have received it within the last 6 months.
* Severe alcoholic hepatitis requiring corticosteroid therapy (Maddrey's Discriminant function ≥ 32 and/or ABIC score > 6.7).
* Patients with active alcohol consumption of more than 21 units per week.
* HIV infection.
* Patients with a history of significant extra hepatic disease with impaired short-term prognosis, including congestive heart failure New York Heart Association Grade III/IV, COPD GOLD >2, chronic kidney disease with serum creatinine >2mg/dL or under renal replacement therapy.
* Patients with current extra hepatic malignancies including solid tumours and hematologic disorders.
* Pregnancy or breastfeeding.
* Patients included in other clinical trials in the month before inclusion.
* Patients with mental incapacity, language barrier, bad social support or any other reason considered by the investigator precluding adequate understanding, cooperation or compliance in the study.
* Refusal to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of ACLF at the end of the study | Month 12

SECONDARY OUTCOMES:
Time to transplant-free survival at months1, 3, 6, 9 and 12 | months 1, 3, 6, 9 and 12
Severity of ACLF assessed by number and types of organ failures at baseline, 1 month, 3 months, 6 months, 9 months and 12 months | months 1, 3, 6, 9 and 12
Frequency of hospital admissions due to complications of cirrhosis assessed at baseline, 1 month, 3 months, 6 months, 9 months and 12 months. | baseline and months 1, 3, 6, 9 and 12
Number of participants developing a new onset episode of ascitis assessed at baseline, 1 month, 3 months, 6 months, 9 months and 12 months | baseline and months 1, 3, 6, 9 and 12
Number of participants presenting worsening of ascitis assessed at baseline, 1 month, 3 months, 6 months, 9 months and 12 months | baseline and months 1, 3, 6, 9 and 12
  Worsening of ascitis will be defined as increased diuretic dosage or need for large-volume parecentesis in patients who had never been treated with this procedure
Percentage of participants developing episodes of renal function impairment assessed at baseline, 1 month, 3 months, 6 months, 9 months and 12 months | baseline and months 1, 3, 6, 9 and 12
  Renal function impairment will be defined by AKI criteria, following criteria of the "EASL Clinical Practice Guidelines for the management of patients with decompensated cirrosis"
Percentage of participants developing the first episode of bleeding by esophageal or gastric varices at baseline, 1 month, 3 months, 6 months, 9 months and 12 months | baseline and months 1, 3, 6, 9 and 12
Number of bleeding episodes by esophageal or gastric varices per patient assessed at baseline, 1 month, 3 months, 6 months, 9 months and 12 months | baseline and months 1, 3, 6, 9 and 12
Number of participants developing a new onset episode of hepatic encephalopathy (HE) assessed at baseline, 1 month, 3 months, 6 months, 9 months and 12 months | baseline and months 1, 3, 6, 9 and 12
Number of participants developing a new onset episode of bacterial infection assessed at baseline, 1 month, 3 months, 6 months, 9 months and 12 months | baseline and months 1, 3, 6, 9 and 12
Changes from baseline in plasma cytokine levels including, but not limited to, TNFα at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in plasma cytokine levels including, but not limited to, IL-6, IL-8, IL-10 and IL-1β at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in plasma cytokine levels including, but not limited to, IFN-ɣ at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in plasma cytokine levels including, but not limited to, G-CSF at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in plasma cytokine levels including, but not limited to, VCAM at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in plasma cytokine levels including, but not limited to, VCAM and VEGF at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in plasma cytokine levels including, but not limited to, oxide form of albumin at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in plasma cytokine levels including, but not limited to, HNA2 at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in plasma cytokine levels including, but not limited to, ADMA and SDMA at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in plasma biomarker FABP4 at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in plasma biomarker sCD-163 at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in plasma biomarker vWF at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in urine biomarker NGAL at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in urine biomarker MCP-1 at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in urine biomarker albumin at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in plasma renin concentration at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in plasma norepinephrine concentration at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in plasma copeptin concentration at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes from baseline in blood levels of bacterial DNA or bacterial products at 3 months, 6 months and 12 months | months 3, 6 and 12
Changes in microbiome composition by analysis of microbial genes and signature at baseline, 3 months, 6 months and 12 months | baseline and months 3, 6 and 12
  The aim of this secondary endpoint is to identify phylogenetic and functional composition in the gut microbiota of patients at different stages of liver disease by analysis of microbial genes and signature.
  As treatment with rifaximin has been associated to changes in microbiota composition in patients with cirrhosis, we will analyze the changes in microbiota signature and composition in patients under treatment with simvastatin and rifaximin at 3 months, 6 months and 12 months
Changes from baseline in liver function evaluated by MELD (Model For End-Stage Liver Disease) score at 1 month, 3 months, 6 months, 9 months and 12 months | months 1, 3, 6, 9 and 12
  MELD score is a system developed to evaluate the severity of chronic liver disease, and it involves serum bilirubin, creatinine and international normalized ratio values
Changes from baseline in liver function evaluated by CLIF-AD (Chronic Liver Failure - Acute Decompensation) score at 1 month, 3 months, 6 months, 9 months and 12 months | months 1, 3, 6, 9 and 12
  CLIF-AD score is a system created to evaluate the prognosis of patients with decompensated cirrosis, and it involves age, white cell count, creatinine, international normalized ratio and sodium
Changes from baseline in liver function evaluated by Child Pugh Score at 1 month, 3 months, 6 months, 9 months and 12 months | months 1, 3, 6, 9 and 12
  Child Pugh is a score created to evaluate the prognosis of patients with cirrosis based on clinical and analytical values. It involves serum bilirubin, coagulation, albumin and the presence of clinical complications of cirrhosis, as hepatic encephalopathy and ascites
Change in quality of life assessed by CLDQ questionnaire (Chronic Liver Disease Questionnaire) at baseline, 1 month, 3 months, 6 months, 9 months and 12 months | baseline and months 1, 3, 6, 9 and 12
  Evaluated by patient administration. CLDQ questionnaire contains 29 items divided into six domains: "Fatigue" which includes perceptions of decreased energy and sleepiness; "Emotional Function" which measures mood and insomnia; "Worry" assessing concerns regarding disease progression and family; "Activity" considering eating habits and movement of heavy objects; and finally, 2 symptom domains, "Abdominal Symptoms" and "Systemic Symptoms". All items refer to the previous 2 weeks on a 7 point Likert scale, with 1 corresponding to the maximum frequency ("all of the time") and 7 to the minimum ("none of the time"). Scores range from 1 (worst) to 7 (least severe), in which higher scores indicate a minimum frequency of symptoms and, consequently, a better quality of life
Change of frailty and functional status assessed by Liver Frailty Index questionnaire at baseline, 1 month, 3 months, 6 months, 9 months and 12 months | baseline and months 1, 3, 6, 9 and 12
  Liver Frailty Index questionnaire is an objectively measure "physical frailty" (a term that we believe embodies these extrahepatic manifestations of cirrhosis) in patients with end-stage liver disease (ESLD) and quantify its impact on health-related outcomes. It's composed by (1) Gender (Male or Female); (2) Dominant hand grip strength (kg), the means of three measures; (3) Chair stands (sec), time that it takes a patient to stand up and sit down in a chair 5 times without using their arms; and (4) Balance (sec), seconds holding 3 position balance tested in 3 positions for 10 seconds each the positions are side by side, semi tandem and tandem.
  Liver Frailty Index is calculated as: (-0:330 * gender-adjusted grip strength) + (-2:529 * number of chair stands per second) + (-0:040 * balance time) + 6.
  The questionnaire does not have a minimum value and a maximum value.
Change of minimal hepatic encephalopathy assessed by PHES questionnaire (Psychometric Hepatic Encephalopathy Score) at baseline, 1 month, 3 months, 6 months, 9 months and 12 months | baseline and months 1, 3, 6, 9 and 12
  The PHES is a questionnaire used in the diagnosis of minimal hepatic encephalopathy (MHE) and can be used to assess motor speed, motor accuracy, concentration, attention, visual perception, visual-spatial orientation, visual construction and memory, which are related to most of neuropsychological impairments in MHE. The PHES is composed of five tests, number connection test-A (NCT-A), number connection test-B (NCT-B), serial dotting test (SDT), line tracing test (LTT) and digit symbol test (DST). This questionnaire measures the time that the patient spends doing the five exercises.
  The questionnaire does not have a minimum value and a maximum value, but as the score increases there is a worsening of outcome.
Changes from baseline in stigmatization assessed by a specific questionnaire at 3 months, 6 months and 12 months | months 3, 6 and 9
  Evaluated by patient administration. This questionnaire quantifies the presence of stigma among patients with cirrhosis. The questionnaire gives a total of 19 stigma-related questions with answer choices based on a four point Likert scale (strongly agree, agree, disagree, and strongly disagree). The questions are divided in four categories 1) discrimination, 2) stereotypes, 3) social isolation and 4) shame. The questionnaire does not have a minimum value and a maximum value, because is only a descriptive questionnaire that values patient perception regarding the disease.
Change in appearance of muscle toxicity at baseline, 1 month, 3 months, 6 months, 9 months and 12 months as defined using a specific statin-associated myopathy questionnaire | baseline and months 1, 3, 6, 9 and 12
  Appearance of muscle toxicity at baseline, 1 month, 3 months, 6 months, 9 months and 12 months as defined using a specific statin-associated myopathy questionnaire. This questionnaire consists of four questions that patients can answer yes or no. The patients met the study definition for "appearance of muscle toxicity" if one of the three of the following occurred: 1) They reported new or increased muscle pain, cramps, or aching, unassociated with exercise; 2) Symptoms persisted for at least 2 weeks; 3) Symptoms resolved within 2 weeks of stopping the study drug; and 4) Symptoms reoccurred within 4 weeks of restarting the study medication.
Number of patients with genetic polymorphisms of statins membrane transporter OATPB1 in all patients included in the study | month 12
Changes from baseline in transaminases at 1 month, 3 months, 6 months, 9 months ans 12 months | months 1, 3, 6, 9 and 12
Changes from baseline in alkaline phosphatase at 1 month, 3 months, 6 months, 9 months ans 12 months | months 1, 3, 6, 9 and 12
Changes from baseline in creatine kinase at 1 month, 3 months, 6 months, 9 months ans 12 months | months 1, 3, 6, 9 and 12
Proportion of patients and severity of treatment-related adverse events during the study period | month 12
Annualized incidence of ACLF during the study period | month 12
Time to overall at the end of the study | month 12
Time to disease related survival at the end of the study | month 12

CONTACTS AND LOCATIONS:
Overall Officials: Pere Ginès, MD, Study Chair — Hospital Clinic of Barcelona
Locations (14):
- University Hospitals Leuven, Leuven, Belgium
- Beajuon Hospital, Clichy, Paris, France
- Universitatsklinikum Frankurt, Frankfurt, Germany
- Italy (3):
  - Bologna University Hospital, Bologna
  - Padova University Hospital, Padua
  - San Giovanni Battista Hospital, Torino
- Academic Medical Centre, Amsterdam, Netherlands
- Spain (6):
  - Hospital Clínic de Barcelona, Barcelona, España
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital de Sant Pau, Barcelona
  - Hospital Moisés Broggi, Barcelona
  - Hospital Parc Taulí, Barcelona
  - Hospital Gregorio Marañón, Madrid
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pose E, Jimenez C, Zaccherini G, Campion D, Piano S, Uschner FE, de Wit K, Roux O, Gananandan K, Laleman W, Sole C, Alonso S, Cuyas B, Ariza X, Juanola A, Ma AT, Napoleone L, Gratacos-Gines J, Tonon M, Pompili E, Sanchez-Delgado J, Allegretti AS, Morales-Ruiz M, Carol M, Perez-Guasch M, Fabrellas N, Pich J, Martell C, Joyera M, Domenech G, Rios J, Torres F, Serra-Burriel M, Hernaez R, Sola E, Graupera I, Watson H, Soriano G, Banares R, Mookerjee RP, Francoz C, Beuers U, Trebicka J, Angeli P, Alessandria C, Caraceni P, Vargas VM, Abraldes JG, Kamath PS, Gines P; LIVERHOPE Consortium. Simvastatin and Rifaximin in Decompensated Cirrhosis: A Randomized Clinical Trial. JAMA. 2025 Mar 11;333(10):864-874. doi: 10.1001/jama.2024.27441. PMID 39908052
- [Derived] Marrache MK, Rockey DC. Statins for treatment of chronic liver disease. Curr Opin Gastroenterol. 2021 May 1;37(3):200-207. doi: 10.1097/MOG.0000000000000716. PMID 33654016